CLINICAL TRIAL: NCT00176293
Title: A Randomized Phase II Trial of Doxil With or Without Dexamethasone in Treatment of Patients With Metastatic Hormone Refractory Prostate Cancer
Brief Title: Randomized Phase II Trial of Doxil With or Without Dexamethasone for Metastatic Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Kentucky (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: John Rinehart, M.D., Principal Investigator, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-GU-52-B
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: prostate; prostate cancer; doxil; dexamethasone; metastatic; hormone refractory
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Dexamethasone; Calcium Dobesilate; Doxorubicin; liposomal doxorubicin

ARMS (2):
- 1 (Experimental): dexamethasone
  Interventions: Drug: dexamethasone; Drug: doxorubicin
- 2 (No Intervention)

INTERVENTIONS:
Drug: dexamethasone — oral dexamethasone, 12mg BID on days 1, 2, 3, 4, & 5 of each 28-day cycle
  Other Names: decadron
  Arms: 1
Drug: doxorubicin — Doxorubicin 50mg/m^2 I.V. on day 5
  Other Names: Doxil
  Arms: 1

SUMMARY:
The primary objective of this study is to assess disease response to Doxil in patients with hormone refractory prostate cancer with or without dexamethasone pre-treatment.

Study Design:

We will perform an open labeled, parallel, randomized phase II study using a two-stage design to determine if there is sufficient anti-tumor activity in either arm to warrant further study. Assumptions made in this study: an unacceptable overall response rate is </= 10% & we will pursue further study if the overall response rate is >/= 30%. Fifteen patients will be randomized in the first phase (to both Arm 1 and Arm 2). No further patients will be accrued if <2/15 responses are noted in a given arm. Ten additional patients will be enrolled if >/= 2/15 responses are observed. If there are >/= 5/25 responses then further studies will be pursued with that regimen. We will determine the overall incidence & severity of toxicities in both arms.

Treatment:

Arm 1: Doxil: Dose: 50 mg/m2, IV (in the vein) on day 5 of each 28 day cycle. Arm 2: Doxil: Dose: 50 mg/m2, IV (in the vein) on day 5 of each 28 day cycle. Arm 1 only: Dexamethasone: Dose: 12 mg twice a day by mouth on days 1, 2, 3, 4, 5 of each 28 day cycle.

Number of Cycles for both Arm 1 & 2: until progression or unacceptable toxicity develops.

DETAILED DESCRIPTION:
Primary Objectives:

To assess the anti-tumor activity of Doxil by assessing response rates in patients with hormone refractory prostate cancer with or without dexamethasone pre-treatment.

Secondary Objectives:

To assess and estimate in patients with hormone refractory prostate cancer treated with Doxil with or without pre-treatment dexamethasone: 1) overall survival 2) toxicity, 3) quality of life parameters, 4) dose intensity administered in both treatment groups.

Study Design:

We will perform an open labeled, parallel, randomized phase II study using a two-stage design to determine if there is sufficient anti-tumor activity in either arm to warrant further study. Assumptions made in this study: an unacceptable overall response rate is </= 10% and we will pursue further study if the overall response rate is >/= 30%. The overall response rate for this study will be based on the total number of responses observed defined as: complete responses + partial responses (both by RECIST)+biochemical responses (in patients with no measurable target lesions a >/= 50% decrease in PSA for >/= 4 weeks). Fifteen patients will be randomized in the first phase (to both Arm 1 and Arm 2). No further patients will be accrued if <2/15 responses are noted in a given arm. Ten additional patients will be enrolled if >/= 2/15 responses are observed. If there are >/= 5/25 responses then further studies will be pursued with that regimen. We will determine the overall incidence and severity of toxicities in both arms.

Treatment:

Arm 1: Doxil: Dose: 50 mg/m2, IV. Frequency: day 5 of each 28 day cycle. Arm 2: Doxil: Dose: 50 mg/m2, IV. Frequency: day 5 of each 28 day cycle. Arm 1 only: Dexamethasone: Dose: 12 mg bid po. Frequency: days 1,2,3,4,5 of each 28 day cycle.

Number of Cycles for both Arm 1 and 2: until progression or unacceptable toxicity develops.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic hormone refractory prostate cancer as defined by resistance to both ablative therapy (with either LHRH agonists or orchiectomy) & anti-androgens.
2. Patients must have symptoms related to disease.
3. Patients must have PS 0,1,2 (ECOG).
4. Patients must have measurable disease (RECIST) or PSA > 5.
5. Patients must have adequate organ function as defined as follows: leukocytes >/= 3,000/mm3, absolute neutrophil count >/= 1,500/mm3, hemoglobin >/= 8.0g/dl, platelets >/= 100,000/mm3, serum creatinine </= 2.5 mg/dl. Bilirubin must be </= 2 fold above ULN. Liver transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional ULN if alkaline phosphatase is </= ULN or alkaline phosphatase may be up to 4 x ULN if transaminases are </= ULN.
6. Patients must have a left ventricular ejection fraction (LVEF) 50% by echocardiogram
7. Patients must have failed to respond to discontinuation of anti-androgens.
8. No previous therapy with anti-androgens, corticosteroids or estrogens in the last 4 weeks.
9. Previous radiation therapy is allowed if completed at least 4 weeks prior to study entry & therapy was cumulatively administered to </= 25% of bone marrow.
10. Patients must be >18 years of age
11. Patients must have an expected survival of at least 4 months.
12. Patients must have the ability to understand & the willingness to sign a written informed consent document.
13. Patients must be willing to use adequate contraceptive method during treatment and for 3 months after completing treatment.

Exclusion Criteria:

1. Patients with previous history of cancer are excluded unless they have had curative treatment completed >/= 5 years prior to entry onto study or had 1 of the following: in situ carcinoma (any location), basal cell carcinoma, or non-metastatic squamous cell carcinoma of the skin.
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, uncontrolled diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements or the ability to provide informed consent.
3. Patients requiring any non study corticosteroids for any reason are excluded.
4. Patients who have received previous chemotherapy.
5. A history of cardiac disease with New York Heart Class II or greater, or clinical evidence of congestive heart failure.
6. Patients may not be receiving any other investigational agents or have participated in any investigational drug study within 4 weeks preceding initiation of treatment.
7. Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from major surgery.
8. Patients with a lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome or inability to swallow tablets.
9. History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL or the components of Doxil®

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with CR or PR | evaluated after 2 courses then every other course

SECONDARY OUTCOMES:
Hematologic toxicity | evaluated @ baseline & 3/wk during treatment or until recovery
Percentage of subjects with >/= Grade 3 hematopoietic & non-hematopoietic toxicities | labs evaluated @ baseline & 3/wk during treatment or until recovery; toxicity evaluated through treatment or until resolved
Clinical non-hematologic & hematologic toxicity | continuous throughout study
QOL | baseline then every other cycle
Fraction delivered vs. intended Doxil | each dose
Cytokines | evaluated days 1, 5, 8 every other cycle
Survival | evaluated through study

CONTACTS AND LOCATIONS:
Overall Officials: John Rinehart, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States